CLINICAL TRIAL: NCT04382612
Title: Assessment of the Safety and Performance of the HARPOON™ Beating Heart Mitral Valve Repair System; a Multi-center Post-market Study (ASCEND)
Brief Title: Treatment of Mitral Regurgitation Using a Minimally Invasive Approach With the HARPOON Device.
Acronym: ASCEND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-22
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HARPOON MVRS (Other): Subjects who were treated with the HARPOON MVRS.
  Interventions: Device: HARPOON Beating Heart Mitral Valve Repair System (MVRS)

INTERVENTIONS:
Device: HARPOON Beating Heart Mitral Valve Repair System (MVRS) — Repair of the chordae tendinae in the mitral valve.

SUMMARY:
To evaluate the long-term safety and performance of the HARPOON™ MVRS for use in patients presenting with severe degenerative mitral regurgitation due to posterior leaflet prolapse in the post-market phase.

DETAILED DESCRIPTION:
This trial is a single arm, prospective, multi-center, non-randomized and open-label post-market study that will evaluate subjects for up to 5 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years old
2. Presence of severe MR as read on a transthoracic echocardiographic study
3. Mitral leaflet coaptation surface is sufficient to reduce mitral regurgitation without undue leaflet tension (approximate leaflet to gap ratio of 2:1) based on the judgment of the patient eligibility committee and the operating surgeon
4. Degenerative mitral valve disease with mid-segment P2 prolapse
5. Patient is able to sign informed consent and able to return for follow-up and is capable of participating in all testing associated with this clinical investigation

Exclusion Criteria:

1. Patient is of the age where further growth is expected
2. Active endocarditis
3. Left ventricular or left atrial appendage thrombus
4. Severe mitral annular and/or leaflet calcification
5. Cannot tolerate procedural anticoagulation or post-procedure antiplatelet regimen
6. Mitral stenosis
7. Functional Mitral Valve disease
8. Previous mitral valve replacement surgery
9. Fragile or thinning apex
10. Contraindications to transoesophageal echocardiography (atlantoaxial disease, severe generalized cervical arthritis, upper gastrointestinal bleeding, significant dysphagia and odynophagia, has received extensive radiation to the mediastinum)
11. Patient is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walther, Prof Dr med, Principal Investigator — Goethe University
Locations (10):
- Austria (2):
  - Medizinische Universität Innsbruck, Universitätsklinik für Herzchirurgie, Innsbruck, Tyrol
  - Kepler Universitätsklinikum GmbH, Linz, Upper Austria
- Germany (6):
  - Universitätsklinik Ulm, Ulm, Baden-Wurttemberg
  - Rhön Klinikum Kardiochirurgie, Bad Neustadt an der Saale, Bavaria
  - Kerckhoff Klinik GmbH, Bad Nauheim, Hesse
  - Schüchtermann Klinik, Bad Rothenfelde, Lower Saxony
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Deutsches Herzzentrum Berlin, Berlin
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands
- Guy's and St Thomas' NHS FOUNDATION TRUST, of Royal Brompton and Harefield Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- HARPOON MVRS: The enrolled cohort with the HARPOON MVRS.
  HARPOON Beating Heart Mitral Valve Repair System (MVRS): Repair of the chordae tendinae in the mitral valve.
Period: Overall Study
Arm/Group | HARPOON MVRS
Started | 42
Completed | 41
Not Completed | 1
Not completed — Screen failure - no attempt to use the device | 1

BASELINE CHARACTERISTICS:
Population: The attempt to treat cohort of the Harpoon MVRS.
Groups:
- HARPOON MVRS: The attempt to treat cohort with the HARPOON MVRS.
  HARPOON Beating Heart Mitral Valve Repair System (MVRS): Repair of the chordae tendinae in the mitral valve.
Arm/Group | HARPOON MVRS
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subject's With Freedom From All-cause Mortality, Disabling Stroke and Life-threatening Bleeding
Description: Subject's freedom from all-cause mortality, disabling stroke and life-threatening bleeding at 30 days post-implant.
Time Frame: 30 days
Population: This outcome is reported as a Kaplan Meier estimate for subjects who were attempted to be treated in the trial where data is available. The number of participants analyzed at the 30-day timepoint is equivalent to the number of patients at risk at that timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | HARPOON MVRS
Number analyzed (Participants) | 38
percentage of subjects | 97.6 [92.8 to 100.0]

2. Primary Outcome: Number of Subjects With Procedural Success During the First 30 Days
Description: Subject's procedural success at 30 days post-treatment, as measured by: Technical success (defined as implantation of at least three chords, leaving the operating room and no conversion to open heart surgery) with reduction of MR to less than or equal to mild and the absence of major device or procedure-related SAEs.
Time Frame: 30 days
Population: Subjects who completed a 30-day follow-up. The outcome is reported for subjects where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | HARPOON MVRS
Number analyzed (Participants) | 38
Participants | 26

ADVERSE EVENTS:
Time Frame: Adverse events occurring from baseline through 24 months post implant of the enrolled cohort.
Groups:
- HARPOON MVRS: The enrolled cohort of the ASCEND trial.
Arm/Group | HARPOON MVRS
All-Cause Mortality (participants affected / at risk) | 1/42
Serious Adverse Events (participants affected / at risk) | 15/42
Other Adverse Events (participants affected / at risk) | 20/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HARPOON MVRS (N=42)
BLEEDING - INTRACARDIAC/INTRATHORACIC INJURY DURING INDEX PROCEDURE (Blood and lymphatic system disorders) | 1 (1)
ARRHYTHMIA - TACHYCARDIA - VENTRICULAR (Cardiac disorders) | 2 (2)
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 1 (1)
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2)
PERICARDITIS (Cardiac disorders) | 1 (1)
REGURGITATION - RECURRENT MITRAL SEVERE (Cardiac disorders) | 5 (5)
DEVICE SPECIFIC COMPLICATION - EPTFE KNOT PULL-OUT/DETACHMENT (FROM LEAFLET) (Product Issues) | 2 (2)
DEVICE SPECIFIC COMPLICATION - OTHER CHORD/KNOT STRUCTURAL PROBLEMS (Product Issues) | 1 (1)
ACUTE KIDNEY INJURY/RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (1)
BONE FRACTURE/BREAK (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER - NONSPECIFIC (General disorders) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (3)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY COMPLICATION - PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HARPOON MVRS (N=42)
ACCESS SITE AND VASCULAR COMPLICATIONS - OTHER MINOR (Vascular disorders) | 1 (1)
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 1 (1)
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 7 (7)
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 1 (1)
ARRHYTHMIA - OTHER (Cardiac disorders) | 1 (1)
REGURGITATION - RECURRENT MITRAL MODERATE (Cardiac disorders) | 1 (1)
REGURGITATION - RECURRENT MITRAL SEVERE (Cardiac disorders) | 1 (1)
DEVICE SPECIFIC COMPLICATION - EPTFE KNOT PULL-OUT/DETACHMENT (FROM LEAFLET) (Product Issues) | 1 (1)
MUSCULAR SKELETAL/DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 2 (2)
NEUROLOGICAL EVENT - TRANSIENT ISCHEMIC ATTACK (TIA) (Cardiac disorders) | 1 (1)
INFECTION/INFLAMMATION - OTHER (Infections and infestations) | 3 (4)
OTHER - NONSPECIFIC (General disorders) | 2 (2)
ALLERGIC REACTION - OTHER (General disorders) | 1 (1)
FEVER - UNKNOWN ORIGIN (General disorders) | 1 (1)
PSYCHIATRIC - OTHER (Psychiatric disorders) | 1 (1)
PSYCHIATRIC DISORDER (Psychiatric disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (5)
RESPIRATORY COMPLICATION - PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY INFECTION - UPPER (URI) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY/RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation to ensure proprietary information shall not be divulged. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT04382612/Prot_SAP_000.pdf